CLINICAL TRIAL: NCT05333861
Title: An Observational, Multicenter Study to Evaluate the Safety and Effectiveness of Hetrombopag in Patients With ITP or AA
Status: Not yet recruiting | Type: Observational
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Collaborators: Jiangsu Hengrui Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: Hetrombopag-ITP/AA
Record Dates: First submitted 2022-04-11; First posted 2022-04-19 (Actual); Last update posted 2022-04-19 (Actual); Status verified 2022-04

CONDITIONS: Primary Immune Thrombocytopenia; Aplastic Anemia
Keywords: Hetrombopag
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic; Anemia, Aplastic | interventions — hetrombopag

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Full-analysis set (FAS): The FAS includes all enrolled patients. The FAS will be used for all analyses.
  Interventions: Drug: hetrombopag

INTERVENTIONS:
Drug: hetrombopag — According to prescription

SUMMARY:
This is a multi-center, observational study in patients with Immune Thrombocytopenia (ITP) or aplastic anemia(AA) designed to describe the real-world safety and effectiveness of hetrombopag and assess the patterns of drug utilization to add to the knowledge base regarding the use of hetrombopag in routine medical practice. Patients eligible for participation will, as part of their routine medical care, be receiving hetrombopag for the treatment of ITP/AA

DETAILED DESCRIPTION:
This is a multi-center, observational study in patients with ITP/AA designed to describe the real-world safety and effectiveness of hetrombopag and assess the patterns of drug utilization to add to the knowledge base regarding the use of hetrombopag in routine medical practice.

Patients eligible for participation will, as part of their routine medical care, be receiving hetrombopag for the treatment of ITP/AA

The scope of the study is to collect both retrospective and prospective data. The main part of the study will be prospective collecting data on usage, effectiveness, safety and patient-reported outcomes whereas the retrospective part will consist of collection of information on previous treatments, reason for treatment switch and, if applicable, hetrombopag treatment prior to enrollment. The retrospective data collection will be based on the information available in the patient's medical records. Data will be collected for up to 12 months prior to hetrombopag treatment start.

Prospective data will be collected at routine clinical visits throughout the study. Patients will be followed for 24 months and will be enrolled until their first scheduled visit after 24 months of enrollment, or until early termination, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

* 1.Established and well documented ITP diagnosis
* 2.Patient is treated with, or at enrollment prescribed hetrombopag for ITP. Decision to initiate treatment shall be made by the treating physician and independently from the decision to include the patient in the study.
* 3.Signed and dated informed consent provided by the patient before any study-related activities are undertaken
* 4.Willing and able to comply with protocol requirements

Exclusion Criteria:

* Enrollment in a concurrent clinical interventional study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The Investigators will attempt to consecutively enroll all eligible patients who present for a routine clinical visit or during a routine visit where the patient is started or continued on hetrombopag treatment
Sampling Method: Non-Probability Sample
Enrollment: 1150 (Estimated)
Dates: Start 2022-05-01 (Estimated); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Adverse events | Data will be collected for all routine visits completed during the study period no more than 24 months.
  Information will be collected via reports from the Investigators based on the patient's medical records and classified according to the National Cancer Institute Common Terminology Criteria for Adverse Events, version 5.0

SECONDARY OUTCOMES:
Number and proportion of patients achieving hematologic response after 3/6/12/24 months treatment | Data will be collected for all routine visits completed during the study period which is no more than 24 months.
  Laboratory measures of CBC will be collected if performed according to routine clinical practice and available in the patient's medical records. All analyses of platelet counts and other hematologic assessments will be based on local laboratory results.
The maximum continuous duration and total duration of response | Data will be collected for all routine visits completed during the study period which is no more than 24 months.
  Hematologic assessments will be based on local laboratory results
Number and proportion of patients requiring rescue medication. | Data will be collected for all routine visits completed during the study period which is no more than 24 months.
  Information will be collected via the patient's medical records.
Change from enrollment in the 36-Item Short Form Survey (SF-36) | Data will be collected for all routine visits completed during the study period which is no more than 24 months.
  SF-36 is a set of generic, coherent, and easily administered quality-of-life measures. These measures rely upon patient self-reporting.
Change from enrollment in the use of concomitant ITP/AA medications throughout the study | Data will be collected for all routine visits completed during the study period which is no more than 24 months.
  Information will be collected via the patient's medical records.
Number and proportion of patients achieving a sustained remission off-treatment (SROT) after discontinuation of hetrombopag | Data will be collected for all routine visits completed during the study period which is no more than 24 months.
  The proportion of responders that were able to taper and discontinue hetrombopag maintaining the response during a period of observation of at least six months.

CONTACTS AND LOCATIONS:
Locations (1):
- Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China